CLINICAL TRIAL: NCT01671306
Title: The Association Between Monocyte Subsets and Coronary Collateral Development in Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ugur ARSLAN, Specialist of Cardiology, Samsun Education and Research Hospital
Other Study IDs: 1037; Samsun EAH (Other: Samsun EAH)
Record Dates: First submitted 2012-08-18; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary collaterals; diabetes mellitus; monocyte subsets
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Collateral, coronary disease: Patients are grouped into 2: Good and poor collateral development
- collateral: Patients are grouped into 2: Good and poor collateral development

SUMMARY:
Monocyte heterogeneity in peripheral blood seems to be important in coronary collateral development in non-diabetic patients with stable coronary artery disease. Our aim in this study is to find out any possible relationship between the levels of circulating monocyte subsets and coronary collateral development in type 2 diabetic patients.

DETAILED DESCRIPTION:
83 diabetic patients with severe coronary artery disease were enrolled in the study. These patients were investigated according to their collateral development. Monocytes and their subtypes, namely CD14++CD16- and CD14+CD16+ cells were compared in 2 groups

ELIGIBILITY:
Inclusion Criteria:

* presence of > 95% stenosis of at least one major coronary artery in their first coronary angiogram.

Exclusion Criteria:

* Patients experiencing acute coronary syndrome either with or without ST elevation in the last one month
* Evidence of ongoing infection and inflammation, known malignancy and chronic kidney disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of 83 consecutive type 2 diabetic patients who have undergone coronary angiography because of stable symptoms and signs of coronary artery disease. The main inclusion criterion was the presence of >95% stenosis of at least one major coronary artery in their first coronary angiogram.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uğur ARSLAN, MD, Principal Investigator — Samsun Education and Research Hospital